CLINICAL TRIAL: NCT04250753
Title: Assessment of Gait Parameters and Their Impact on Postoperative Recovery in Patients with Lumbar Spinal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-2019-claudication
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: neurogenic claudication; gait parameters; walking impairment
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with lumbar spinal stenosis
  Interventions: Other: Walking task

INTERVENTIONS:
Other: Walking task — 30 meters walking task (15 meters round trip) following by a rest period of 2 minutes. Participants are invited to perform the 30 meters walking task twice. Inertial sensors are put on each participant foot.

SUMMARY:
The objective is to observe the evolution of walking parameters during the surgery process and find which of all calculated walking parameters represent the best indicators of functional disabilities and postoperative recovery for patient with lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar spinal stenosis
* Presenting neurogenic claudication
* Waiting for a surgery (laminectomy, laminotomy, fusion)

Exclusion Criteria:

* Symptomatic hip or knee osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old with lumbar spinal stensois
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline French-Canadian adaptation of Swiss Spinal Stenosis Questionnaires (FC-SSSQ) | Baseline, 6 weeks post-surgery, 6 months post-surgery
  pain, function and satisfaction related to lumbar spinal stenosis. Pain subscale score range from 7 to 35 with higher values indicate a worst outcome, Function subscale score range from 5 to 20 with higher values indicate a worst outcome, Satisfaction subscale score range from 6 to 24 with higher values indicate a worst outcome. The total score is composed of the three subscales and range from 18 to 79.
Change from baseline Quality of life (EuroQol - 5D) | Baseline, 6 weeks post-surgery, 6 months post-surgery
  Quality of life related to mobility, self-care, usual activities, pain and discomfort, anxiety and depression. Each category has a score ranging from 1 to 3 and higher values indicate a worst outcome.
Change from baseline International Physical Activity Questionnaire (IPAQ) | Baseline, 6 weeks post-surgery, 6 months post-surgery
  physical activity habits. IPAQ score range from 1 to 3 where a score of 3 indicates a higher practice of physical activity
Change from baseline Walking time | Baseline, 6 weeks post-surgery
  Time participants take to do the walking task in seconds
Change from baseline Walking speed | Baseline, 6 weeks post-surgery
  the walking stride velocity (meter/second) is the mean speed of forward walking, calculated in meters per second
Change from baseline Gait cycle | Baseline, 6 weeks post-surgery
  Gait cycle (% stance phase, % swing phase)
Change from baseline Stride length | Baseline, 6 weeks post-surgery
  Stride Length [m] describes the distance between two successive footprints on the ground, from the heel of a foot to the heel of the same foot, one cycle after.

SECONDARY OUTCOMES:
Change from baseline Swing Width | Baseline, 6 weeks post-surgery
  Swing Width (m) is the maximal lateral excursion of the foot during swing phase. It is the maximum lateral distance between the forward path and the real path of the foot.
Change from baseline Minimal To Clearance | Baseline, 6 weeks post-surgery
  Min. Toe Clearance (meter) is the minimum height of the toes during swing phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada